CLINICAL TRIAL: NCT03339531
Title: Definition of Fields Margins for Optimized 2D Radiotherapy of Prostate Carcinoma
Brief Title: Optimized 2D-RT for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2D-RT in prostate cancer
Record Dates: First submitted 2017-11-03; First posted 2017-11-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
Keywords: 2D; prostate neoplasms; radiotherapy; simulation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2D radiotherapy (Experimental): Patients with prostate cancer were treated with 2D-radiotherapy
  Interventions: Radiation: 2D radiotherapy

INTERVENTIONS:
Radiation: 2D radiotherapy

SUMMARY:
Prostate cancer (CAP) is one of the most common malignancies in men, both in Western countries and developing countries. Radiation therapy (RT) is an important therapeutic option. New technologies (3D, IMRT, IGRT, VMAT) have been introduced in the last decades, with a progressive improvement of clinical outcome. However, in many countries the only treatment option is the traditional 2D technique based on standard simulation. The indications for field definition in this treatment are still based on expert's opinions. The aim of this analysis is to propose new indications for 2D fields definition based on three-dimensional simulation in a population of patients with CAP. Twenty patients with CAP consecutively treated with RT in our center were identified. Patients underwent CT-simulation in supine position. Pelvic MRI images were fused with CT-simulation images. In this way, delineation of the prostate and seminal vesicles was performed on MRI images. Clinical Target Volume definition (CTV) was performed according to EORTC guidelines simulating 4 different categories: low-risk CAP, intermediate-risk CAP, high-risk CAP without involvement of the seminal vesicles, and high-risk CAP with involvement of seminal vesicles. The Planning Target Volume (PTV) was defined by adding a margin of 10 mm to the CTV in all directions. For each patient, 8 treatment plans were calculated. In particular, for each of the 4 categories of risk, 2 treatment plans were calculated by using a cobalt source or 10 MV photons. Treatment plans were calculated using the box technique. Progressive optimization was realized with an iterative procedure by evaluating the three-dimensional dose distribution. Once the final plan was achieved (respecting the PTV constraint: D98 > 95%), distances of the fields edges from a set of reference points were measured.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* clinical T stage: cT2b, cT2c, cT3a, cT3b
* informed consent
* MRI of the pelvis

Exclusion Criteria:

* > 79 years
* prior surgery treatment for prostate cancer
* prior pelvic radiotherapy
* genetic syndromes of hyper-radio-sensitivity
* chronic infiammatory bowel disease

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
new indications for 2D fields definition | through study completion, up to 10 months
  Twenty patients with prostate cancer (CAP) were identified. Pelvic MRI images were fused with CT-simulation images to delineate prostate and seminal vesicles on MRI images. Clinical Target Volume definition (CTV) was performed according to EORTC guidelines simulating 4 different categories: low-risk CAP, intermediate-risk CAP, high-risk CAP with or without involvement of the seminal vesicles. The Planning Target Volume (PTV) was defined by adding a margin of 10 mm to the CTV. For each patient, 8 treatment plans were calculated using box tecnhique: 2 treatment plans for each risk category were calculated by using a cobalt source or 10 MV photons. Progressive optimization was realized with an iterative procedure by evaluating the three-dimensional dose distribution. Once the final plan was achieved (respecting the PTV constraint: D98 > 95%), distances of the fields edges from a set of reference points were measured.

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, MD, Study Director — Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine-DIMES, Unversity of Bologna, S. Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No